CLINICAL TRIAL: NCT01930955
Title: Non-antibiotic Prescribing for Acute Upper Respiratory Tract Infection：a Randomized-control Trial
Brief Title: Non-antibiotic Prescribing for Acute Upper Respiratory Tract Infection
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no patients were included
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, Chen Long,MD, Prof;MD, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AURI
Record Dates: First submitted 2013-08-20; First posted 2013-08-29 (Estimated); Last update posted 2023-05-01 (Actual); Status verified 2021-02

CONDITIONS: Acute Upper Respiratory Tract Infection
Keywords: Non-antibiotic prescribing; acute upper respiratory tract infection; white cell count; vomiting
MeSH Terms: conditions — Vomiting | interventions — Amoxicillin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Amoxicillin (Active Comparator): Amoxicillin were given to the children with acute upper respiratory tract infection characterized by fever and vomiting.
  Interventions: Drug: Amoxicillin
- control (No Intervention): Non-antibiotics were given to the children with acute upper respiratory tract infection characterized by fever and vomiting.

INTERVENTIONS:
Drug: Amoxicillin — β-lactam antibiotics
  Arms: Amoxicillin

SUMMARY:
Some acute upper respiratory tract infection(AURI) in children is characterized by fever and vomiting,and it is one common reason for visiting a pediatrician. White blood count(WBC) usually increased in this children patients,hence antibiotics are often prescribed properly assumed. In the present study, it was hypothesized that it was not necessary to prescribe amoxicillin for the children.

DETAILED DESCRIPTION:
After inclusion of eligible children patients,one group was prescribed amoxicillin,and another not.

ELIGIBILITY:
Inclusion Criteria:

* Acute upper respiratory tract infection
* Fever
* Vomiting
* Increased white blood cell

Exclusion Criteria:

* 0ther symptoms of digestive system
* Headache

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2011-08-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
fever | 3 days
  Fever stopped or mitigated in 90% participants.

SECONDARY OUTCOMES:
vomiting | 2 days
  Vomiting stopped or mitigated in 90% participants.

OTHER OUTCOMES:
white cell count | 3 days
  White cell count decreased in 90% participants.

CONTACTS AND LOCATIONS:
Overall Officials: Long Chen, MD, Principal Investigator — Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Locations (1):
- Department of Pediatrics, Daping Hospital, Research Institute of Surgery, Third Military Medical University, Chongqing, Chongqing Municipality, China